CLINICAL TRIAL: NCT07359157
Title: Changing Lives and Changing Outcomes-9 at Worcester Recovery Center and Hospital: Implementing and Evaluating A Mental Illness and Criminal Risk Focused Intervention for People With Serious Mental Illness
Brief Title: Changing Lives and Changing Outcomes-9 at Worcester Recovery Center and Hospital
Acronym: CLCO-9
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Worcester Recovery Center and Hospital (Unknown)
Responsible Party: Principal Investigator, Faith Scanlon, Counseling Psychologist, Instructor of Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000801
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Serious Mental Illness; Psychotic Disorder; Depression; Bipolar
Keywords: serious mental illness; criminogenic risk; criminal legal involvement; treatment; forensic; state hospital
MeSH Terms: conditions — Psychotic Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Changing Lives and Changing Outcomes-9 Group (Experimental): Changing Lives and Changing Outcomes-9, a brief cognitive-behavioral therapy intervention for people with mental illness involved in the legal system, will be administered in treatment groups consistent with standard programming at the state hospital. Patients will be able to participate in this group in addition to any other services at the hospital.
  Interventions: Behavioral: Changing Lives and Changing Outcomes-9

INTERVENTIONS:
Behavioral: Changing Lives and Changing Outcomes-9 — A brief, cognitive therapy-based intervention for people with mental illness and legal system involvement.
  Other Names: CLCO-9

SUMMARY:
People with serious mental illness (depression, bipolar, and schizophrenia spectrum disorders) have high rates of repeated criminal legal involvement and psychiatric hospitalizations. Longstanding research shows that in addition to treating clients' symptoms of mental illness, targeting risk factors for legal involvement can help reduce their chances of future incarcerations. Because hospitals are becoming increasingly forensic, treatment programs that address both mental illness and risk factors for legal involvement may be especially helpful in a state hospital setting, like Worcester Recovery Center and Hospital (WRCH). This treatment study offers an adjunctive 9-session intervention, Changing Lives and Changing Outcomes-9 (CLCO-9), for patients at WRCH; this program is designed to help people with serious mental illness who are involved in the legal system increase their awareness of their mental health and reduce their chances of future legal involvement.

The investigators are proposing a treatment study testing the use of the CLCO-9 group intervention with patients with serious mental illness with current or previous criminal legal involvement at Worcester Recovery Center and Hospital (WRCH). The study has three aims:

1. Evaluate feasibility, fidelity, and patient satisfaction during the implementation of the CLCO-9 group treatment at WRCH
2. Evaluate CLCO-9's effectiveness on improving patient's self-reported mental health, and behavioral indicators of mental health and risk factors for legal involvement
3. Explore changes in WRCH clinicians' knowledge and attitudes about treating risk factors for criminal legal involvement.

To test these aims, the research team will employ a two-phase study. In the first phase, the researchers will implement the intervention and make necessary adjustments to maximize the success of the implementation. In the second phase, the researchers will evaluate the treatment program's effectiveness in producing change from pre- to post-treatment.

All patient participants in this study will receive the intervention. The projected sample size is about 20 treatment completers and 4 to 8 group leaders.

DETAILED DESCRIPTION:
In this treatment study, the investigators propose to implement and evaluate a 9-session intervention, cognitive-behavioral intervention, Changing Lives and Changing Outcomes-9 (CLCO-9), for patients at Worcester Recovery Center and Hospital (WRCH) with serious mental illness (i.e., depression, bipolar, and psychotic disorders) with current or previous legal involvement.

The CLCO-9 groups will be led by WRCH clinical staff/trainees who have competed a clinical training in the CLCO-9 intervention led by Dr. Scanlon (PI). This study is comprised of two parts: a clinical phase, and then the effectiveness phase (see Section 5.7 Study Procedures). The study is guided by the following aims:

Aim 1 will evaluate feasibility, fidelity, and patient satisfaction during the implementation of the CLCO-9 group treatment at WRCH.

The researchers hypothesize the implementation will demonstrate feasibility based on the number of patients who agree to join the group and attendance. The researchers anticipate approximately 40 patients will agree to participate in the study, with a projected sample size of 20 treatment completers (i.e., patient participants who attended 5 or more of the 9 group sessions and post-treatment measures). Using transcriptions from consultation calls with group leaders on clinical and implementation issues, the research team will also explore barriers and facilitators of the intervention's feasibility.

The researchers hypothesize that group leader participants will report high levels of session fidelity to the treatment program per session fidelity checklists (i.e., ≥ 75% of session content covered, on average, per session).

The researchers hypothesize patient participants will report satisfaction with CLCO-9 treatment sessions (per the Client Satisfaction Questionnare-8).

The researchers will also explore patient engagement in each session, per group leader participant report on a scale of 1 (disengaged) to 5 (exemplary). The research team will collect patients' session homework to explore homework completion as another indicator of engagement.

Aim 2 will evaluate the CLCO-9's effectiveness in improving patient-reported and behavioral indicators of mental health and criminal risk.

From pre-to post-treatment, the researchers hypothesize improvements in patient-reported emotional distress (per the Modified Colorado Symptom Index), aggression and hostility (per the Bus-Perry Aggression Questionnaire), criminal thinking (per the Psychological Inventory of Criminal Thinking Styles-Short Form), antisocial attitudes (per the Measure of Criminal Attitudes and Associates Part B), and knowledge of treatment content (per the CLCO-9 knowledge quiz) will improve from pre- to post-treatment.

The investigators hypothesize that, per WRCH chart review, behavioral outcomes will show reduced Broset Violence Checklist scores and fewer restraints/seclusions from before to immediately after treatment. The research team also hypothesizes treatment recipients will show improved treatment engagement (i.e., attending more treatment meetings and other groups) across treatment.

Aim 3 will evaluate the changes in WRCH CLCO-9 clinician knowledge and attitudes about treating criminal risk.

The investigators hypothesize that clinicians will show increased knowledge (per the Knowledge about Addressing Criminal Risk quiz) and attitudes (per the Staff Responses to Attitude scale) on addressing criminal risk among patients with SMI after leading the CLCO-9 groups. Change will be calculated by comparing pre-training survey data, post-training survey data, and follow-up survey data after group leaders complete their first and last groups.

ELIGIBILITY:
Inclusion Criteria:

* Currently hospitalized at Worcester Recovery Center and Hospital (WRCH)
* At least 18 years old
* Self-reported current or past legal involvement
* Speaks English
* For patients without a legally authorized representative (LAR): demonstrate capacity to consent per the Capacity Assessment Record (CAR).
* For patients with an LAR: assent to participate.

Exclusion Criteria:

* Hospital status that does not permit group attendance (e.g., room-based seclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Buss-Perry Aggression Questionnaire | From before starting treatment (baseline assessment) to after completing treatment (anticipated to be about 7 weeks after starting treatment)
  aggression and hostility
Modified Colorado Symptom Index | From before starting treatment (baseline assessment) to after completing treatment (anticipated to be about 7 weeks after starting treatment)
  emotional distress
Psychological Inventory of Criminal Thinking Styles-Short Form | From before starting treatment (baseline assessment) to after completing treatment (anticipated to be about 7 weeks after starting treatment)
  criminal thinking
Measure of Criminal Attitudes and Associates | From before starting treatment (baseline assessment) to after completing treatment (anticipated to be about 7 weeks after starting treatment)
  antisocial attitudes
CLCO-9 knowledge quiz | From before starting treatment (baseline assessment) to after completing treatment (anticipated to be about 7 weeks after starting treatment)
  treatment content

SECONDARY OUTCOMES:
Feasibility of implementation | From patient recruitment until study ends (anticipated to be about 6 months after recruitment begins)
  number of patients who agree to join the group and attendance
Treatment fidelity | Measures after each session for the duration of treatment offered as part of the study (anticipated: about 6 months from recruitment start to study end)
  Session fidelity to the CLCO-9 treatment program (per session fidelity checklists)
Client Satisfaction Questionnare-8 | After each session for the duration of treatment offered during the study (anticipated to be about 6 months)
  Patient satisfaction
Broset Violence Checklist scores | One month before starting treatment to after completing study, which is anticipated to be about 7 weeks after baseline (e.g., after completing post-treatment assessments or discharge, whichever comes first).
  Behavioral indicator documented in patient chart as a staff-rated indicator of imminent patient violence (only available if patient gives permission for chart review)
Patient restraint/seclusion events | One month before starting treatment to after completing study, which is anticipated to be about 7 weeks after baseline (e.g., after completing post-treatment assessments or discharge, whichever comes first).
  Behavioral indicator documented in patient chart of instances that patient was restrained/secluded during current hospitalization (only available if patient gives permission for chart review)
Patient engagement in other treatment meetings/groups | One month before starting treatment to after completing study, which is anticipated to be about 7 weeks after baseline (e.g., after completing post-treatment assessments or discharge, whichever comes first).
  Behavioral indicator documented in patient chart of patient's engagement in treatment meetings and groups beyond the CLCO-9 group during the current hospitalization (only available if patient gives permission for chart review)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Scanlon, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Worcester Recovery Center and Hospital, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not have a plan to share individual participant data with other researchers.